CLINICAL TRIAL: NCT02542735
Title: Incidence of Type 2 Diabetes in the di@Bet.es Study: Role of Fatty Acid Transport System Regulated by VEGFB in the Development of Metabolic Diseases.
Brief Title: Incidence of Type 2 Diabetes in the di@Bet.es Study
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Spanish Biomedical Research Centre in Diabetes and Associated Metabolic Disorders (Other)
Responsible Party: Principal Investigator, Gemma Rojo, Senior Researcher, Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud
Other Study IDs: PI14/00710
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Serum and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spanish di@bet.es cohort: Representative of Spanish population

SUMMARY:
Our aim was to determine the incidence of type 2 diabetes mellitus in a nation-wide population based cohort from Spain (di@bet.es study). The target was the Spanish population. The sample consisted of 5072 people older than 18 years, in 100 clusters (health centres randomly selected from all over Spain). The following variables were recorded: Socio-demographic and clinical data, survey on habits (physical activity and frequency of selected food consumption) and a physical examination was made (weight, height, waist, hip, blood pressure). A fasting blood draw and an oral glucose tolerance test were performed. Determinations of serum glucose were made. In the follow-up the same variables were collected and HbA1c was determined. A total of 2408 subjects participated in the follow-up (7.5±0.6 years, 39.7% men). In total, 154 people developed diabetes (6.4% cumulative incidence in the 7.5 years of follow-up). The incidence of total diabetes adjusted for the structure of age and sex of the Spanish population was 11.6 cases/1000 person-years (IC95%=11.1-12.1). The incidence of known diabetes was 3.7 cases/1000 person-years (IC95%=2.8-4.6) and the incidence of unknown diabetes was 7.9 cases/1000 person-years (IC95%=5.3-8.1). The main risk factors for developing diabetes were the presence of prediabetes in cross-sectional study, age, male sex, obesity, central obesity, increase in weight, and family history of diabetes. This work provides data about population-based incidence rates of diabetes and associated risk factors in a nation-wide cohort of Spanish population.

ELIGIBILITY:
Inclusion Criteria:

* General Population

Exclusion Criteria:

* diabetes in cross-sectional study
* serious illness that prevents participation
* pregnancy
* surgery within the previous month
* any other disabling situation that prevents participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is based on the di@bet.es study, a cross-sectional study undertaken from 2007-2010 from a random cluster sampling in the Spanish population over 18 years of age (Soriguer et al. Diabetologia 2012;55(1):88-93).
Sampling Method: Probability Sample
Enrollment: 2408 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Type 2 diabetes incidence | 6 years on average
  Presence of type 2 diabetes mellitus diagnosed by OGTT after 6 years of follow up in a Spanish population.
Metabolic syndrome incidence | 6 years on average
  Presence of metabolic syndrome (according ATPIII criteria) after 6 years of follow up in a Spanish population.

SECONDARY OUTCOMES:
Risk of diabetes according to each of the measured SNP | 6 years on average
  To show that the presence of particular alleles of genes encoding fatty acid transporters and their regulatory proteins (VEGF-B) are associated with the risk of developing type 2 diabetes after six years of follow up.
Risk of metabolic syndrome according to each of the measured SNP | 6 years on average
  To show that the presence of particular alleles of genes encoding fatty acid transporters and their regulatory proteins (VEGF-B) are associated with the risk of developing metabolic syndrome after six years of follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Universitario, Málaga, Malaga, Spain

REFERENCES:
- [Background] Soriguer F, Goday A, Bosch-Comas A, Bordiu E, Calle-Pascual A, Carmena R, Casamitjana R, Castano L, Castell C, Catala M, Delgado E, Franch J, Gaztambide S, Girbes J, Gomis R, Gutierrez G, Lopez-Alba A, Martinez-Larrad MT, Menendez E, Mora-Peces I, Ortega E, Pascual-Manich G, Rojo-Martinez G, Serrano-Rios M, Valdes S, Vazquez JA, Vendrell J. Prevalence of diabetes mellitus and impaired glucose regulation in Spain: the Di@bet.es Study. Diabetologia. 2012 Jan;55(1):88-93. doi: 10.1007/s00125-011-2336-9. Epub 2011 Oct 11. PMID 21987347